CLINICAL TRIAL: NCT04758039
Title: Clinical Characteristics and In-hospital Death During the First 100 Days of the COVID-19 Pandemic in Chile: A Prospective Cohort Study From a University Hospital
Brief Title: Clinical Characteristics and In-hospital Death of a Chilean COVID-19 Prospective Cohort
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Francisco Gonzalez, Assistant Professor, University of Chile
Other Study IDs: OAIC N° 1119/20
Record Dates: First submitted 2021-02-15; First posted 2021-02-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Corona Virus Infection
Keywords: Coronavirus Infection; COVID-19; SARS-CoV 2; Clinical Scenarios; Hospitalism; Hospitalist; Teaching Hospital; Awake Prone Positioning; Ventilated Prone Positioning; High Flow Nasal Cannula; HFNC; Invasive Mechanical Ventilation; Modified Charlson Comorbidity Index; Charlson Comorbidity Index; In-Hospital Mortality
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators planned to examine a cohort of admitted patients at University of Chile Clinical Hospital with COVID-19 diagnosis. Authors report data on mortality, ICU admission, need of invasive mechanical ventilation, awake and ventilated prone positioning, use of High Flow Nasal Cannula, Thromboembolic disease, Acute Kidney Injury (AKI) and Renal Replacement Therapy. Additionally, the risk of in-hospital death according to chronic disease burden and severity of illness at admission was assessed.

DETAILED DESCRIPTION:
This is a prospective cohort study of adult inpatients at University of Chile Clinical Hospital, located in Santiago, Chile. We enrolled all patients aged over 18 years detected with COVID-19 admitted to the emergency department between March 1-June 11, 2020 through prospective identification using daily admission records. Briefly, COVID-19 diagnosis was made when patients had clinical findings of acute respiratory illness together with i) a positive result on reverse transcriptase chain reaction polymerase (RT-PCR) assay performed on a nasopharyngeal swab; and/or ii) chest computed tomography (CT) with typical findings of COVID-19 and absence of an alternative diagnosis. We intended to include all admitted patients during the first 100 days of the pandemic; therefore, no sample size calculation was performed. We excluded patients with length of stay less than 24 hours, nosocomial SARS-CoV-2 infection, and asymptomatic patients admitted for causes unrelated to SARS-CoV-2 infection regardless of their admission RT-PCR result.

All data were prospectively recorded for each included patient at admission and then daily until the end of the follow-up. Records were consulted by trained physicians, using a standardized data collection form, and then checked by a team of four physicians. Data discrepancy was agreed between the same clinicians.

Recorded data included demographic characteristics, comorbidities, disease onset time, associated symptoms, vital signs at the emergency department, laboratory test performed within 24 hours after admission, characteristics of the first chest CT, medication and supportive care provided, and length of stay at the hospital.

The use of antibiotics, antiviral therapy, corticosteroids, advanced oxygen delivery techniques, need for invasive mechanical ventilation (IMV), awake and ventilated prone position, use of vasopressor drugs, and need for renal replacement therapy (RRT) were explicitly recorded. Clinical management and use of these therapies were based on national recommendations from scientific societies and local protocols. Outcome collection and assignment are explained below.

Laboratory confirmation of SARS-CoV-2 infection was made using RT-PCR of nasopharyngeal swabs. All laboratory, microbiologic, and radiologic assessments were performed at the discretion of the treating physicians who were encouraged to follow local clinical guidelines. Film-array on the nasopharyngeal swab was performed for viral co-infection assessment, and urinary antigens. (pneumococcal and legionella) and blood cultures were performed for bacterial co-infection assessment. Chest radiographs and CT were also performed for all inpatients by experienced radiologists and classified as COVID-19-unrelated, typical or atypical pattern, and unspecified.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Diagnosis of COVID-19 defined by clinical findings of acute respiratory illness (as per WHO guidelines) together with i) a positive result on reverse transcriptase chain reaction polymerase (RT-PCR) assay performed on a nasopharyngeal swab; and/or ii) chest computed tomography (CT) with typical findings of COVID-19 and absence of an alternative diagnosis

Exclusion Criteria:

* Length of hospital stay less than 24 hours
* Nosocomial SARS-CoV-2 infection
* Asymptomatic patients admitted for causes not related to coronavirus infection regardless their admission RT-PCR result

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with confirmed infection by SARS-CoV 2 Since the purpose of this study was to include all the patients admitted during the first 100 days of the pandemic, no sample size calculation was performed.
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
In hospital Mortality | March 13th to July 10th 2020
  Death while hospitalized

SECONDARY OUTCOMES:
Admission to an intensive care unit (ICU) | March 13th to July 10th 2020
  Admission to an intensive care unit (ICU)
Use of invasive mechanical ventilation (IMV) | March 13th to July 10th 2020
  Days from admission and length of IMV
Presence of thromboembolic disease (deep vein thrombosis, pulmonary embolism or both) | March 13th to July 10th 2020
  Described as a positive US exploration of the arms or legs, and a positive CT Scan
Acute kidney injury (AKI) | March 13th to July 10th 2020
  AKI, as per defined by the Kidney Disease Improving Global Outcomes (KDIGO) initiative
Renal replacement therapy (RRT). | March 13th to July 10th 2020
  Days from admission and length of RRT

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Gonzalez, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clinico de la Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be shared upon request